CLINICAL TRIAL: NCT02478320
Title: A Proof-of-Concept Study for Ilorasertib (ABT-348) Activity in Patients With CDKN2A-Deficient Advanced Solid Cancers: a Phase II Basket Trial
Brief Title: Phase II Study of Ilorasertib (ABT348) in Patients With CDKN2A Deficient Solid Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to company's decision to discontinue drug development
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0920; NCI-2015-01251 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-06-19; First posted 2015-06-23 (Estimated); Results first posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Advanced Cancers
Keywords: Advanced Cancers; CDKN2A-Deficient Advanced Solid Cancers; Advanced or metastatic cancer.; Ilorasertib; ABT-348
MeSH Terms: conditions — Neoplasm Metastasis | interventions — ilorasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ilorasertib (ABT-348) (Experimental): Part 1 Dose of Ilorasertib: 200 mg administered by mouth twice daily on Days 1, 8, and 15 of each 28-day cycle.
  Part 2 Expansion: Ilorasertib200 mg administered by mouth twice daily on Days 1, 8, and 15 of each 28-day cycle.
  Interventions: Drug: Ilorasertib

INTERVENTIONS:
Drug: Ilorasertib — 200 mg administered by mouth twice daily on Days 1, 8, and 15 of each 28-day cycle.
  Other Names: ABT-348

SUMMARY:
The goal of this clinical research study is to learn if ilorasertib (ABT-348) can help to control CDKN2A-deficient cancer. CDKN2A deficiency is a type of mutation (a genetic change). The safety of this drug will also be studied.

DETAILED DESCRIPTION:
Study Drug Administration:

Each study cycle is 28 days. You will take ABT-348 by mouth 2 times each day on Days 1, 8, and 15 of each cycle. The first dose you take on these days is called Dose 1, and the second dose you take each day is called Dose 2.

You will take Dose 1 (the earlier dose) of ABT-348 with 4 ounces (about ½ cup) of water. You should fast (not eat or drink anything except water) for 8 hours before taking this dose. You need to fast before this dose because eating food may affect the levels of the study drug that is able to enter your system. You will be allowed to have a light snack 2 hours after Dose 1, and then you may eat anything you like 4 hours after the dose.

You should take Dose 2 (the later dose) as close as possible to 6 hours after the first dose, but not less than 6 hours after the first dose. You do not need to fast before Dose 2. You may eat and drink normally around this dose.

Study Visits:

On Day 1 of each cycle, and on Days 8 and 15 of Cycles 1 and 2:

* You will have a physical exam.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* You will have an EKG (Day 1 of Cycle 2 only). For Cycle 3 and after, you will have these EKGs repeated every 3 cycles (Cycles 6, 9, 12, and so on).

On Day 1 of all cycles, urine will be collected for routine tests.

On Day 1 of Cycles 2 and beyond, if you can become pregnant, blood (about 1 teaspoon) or urine will be collected for a pregnancy test.

Every 8 weeks, you will have a chest x-ray, bone scan, MRI/CT or PET/CT to check the status of the disease.

You may be able to have some of these tests/procedures performed at a local lab, clinic, or doctor's office that is closer to your home. The results of these tests will be sent to the study doctor for review. The study doctor or research staff will discuss this option with you in more detail.

Length of Study Drug Administration:

You may continue taking the study drug for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

You participation on this study will be over after your last dose of study drug.

This is an investigational study. ABT-348 is not FDA approved or commercially available. It is currently being used for research purposes only. The study doctor can explain how the study drug is designed to work.

Up to 65 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed, advanced or metastatic cancer for which standard curative or palliative measures do not exist or are no longer effective.
2. Patients must have CDKN2A-deficient tumor (deletion or mutation). Definition of CDKN2A deficient tumor: #1. CDKN2A deletion or mutation by any CLIA-certified sequencing OR #2. >/= 30% of tumor cells with (at least) hemizygous deletion by FISH. Status will be determined from archived tissue.
3. Patients must have measurable disease by RECIST 1.1.
4. Patients must be >/=18 years of age.
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2.
6. Subject has adequate renal function as demonstrated by serum creatinine value of </= 1.5 times the upper limit of normal (ULN) and either an estimated creatinine clearance value of >/= 50 mL/min as determined by the Cockcroft-Gault formula or a creatinine clearance value of >/= 50 mL/min based on a 24 hour urine collection.
7. Subject has adequate liver function as demonstrated by serum bilirubin </= 2 x ULN and AST and ALT </= 2.5 x ULN. For subjects with liver metastasis, adequate liver function is demonstrated by serum bilirubin </= 2 x ULN and AST/ALT </= 5.0 x ULN.
8. Subject has adequate bone marrow as demonstrated by absolute neutrophil count (ANC) >/= 1,500/mm3 (1.5 x 10^9/L); Platelets >/= 100,000/mm2 (100 x 10^9/L); Hemoglobin >/= 9.0 g/dL (1.4 mmol/L).
9. Subject has QTc interval < 500 msec on baseline electrocardiogram.
10. The subject has a documented Left Ventricular Ejection Fraction > 50%.
11. Women of child-bearing potential and men must agree to use adequate contraception (one of the following listed below) prior to the study entry, for the duration of study participation and up to 3 months following completion of therapy. Women of child-bearing potential must have a negative pregnancy test within 7 days prior to initiation of treatment and/or post menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. -Total abstinence from sexual intercourse (minimum one complete menstrual cycle) -Vasectomized male subjects or vasectomized partner of female subjects -Intrauterine device -Double-barrier method (condoms, contraceptive sponge, diaphragm or vaginal ring with spermicidal jellies or cream) -Additionally, male subjects (including those who are vasectomized) whose partners are pregnant or might be pregnant must agree to use condoms for the duration of the study and for 3 months following completion of therapy.
12. Ability to understand and willingness to sign informed consent form prior to initiation of the study and any study procedures.
13. Signed informed consent approved by the Institutional Review Board prior to patient entry

Exclusion Criteria:

1. Patients with CDKN2A wild type by a CLIA-certified laboratory
2. Subject has known active CNS involvement. The subject has untreated brain or meningeal metastases. CT scans are not required to rule out brain or meningeal metastases unless there is a clinical suspicion of central nervous system disease. Subjects with treated brain metastases that are radiographically or clinically stable for at least 4 weeks after therapy and have no evidence of cavitation or hemorrhage in the brain lesion(s) are eligible, providing that they are asymptomatic, and do not require corticosteroids (must have discontinued steroids at least 1 week prior to study drug administration).
3. Subject has received anti-cancer therapy including chemotherapy, immunotherapy, radiotherapy, hormonal, biologic or any investigational therapy within a period of 21 days or 5 half-lives (whichever is shorter) prior to Study Day 1.
4. Subject has unresolved toxicities from prior anti-cancer therapy, defined as any Common Terminology Criteria for Adverse Events (NCI CTCAE v 4.0) grade 2 or higher clinically significant toxicity (excluding alopecia).
5. Subject has had major surgery within 28 days prior to Study Day 1.
6. Subject currently exhibits symptomatic or persistent, uncontrolled hypertension defined as diastolic blood pressure > 90 mmHg or systolic blood pressure > 140 mmHg. Subjects may be re-screened if blood pressure is shown to be controlled with or without intervention.
7. Subject has proteinuria defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v 4.0) grade > 1 at baseline as measured by a urine dipstick (2+ or greater) and confirmed by a 24 hour urine collection (>/= 1 g/24 hrs). Subjects may be re-screened if proteinuria is shown to be controlled with or without intervention.
8. Subject is receiving therapeutic anticoagulation therapy. Low dose anti-coagulation (e.g., low dose heparin or warfarin) for catheter prophylaxis will be permitted. Use of Aspirin for treatment of Atrial Fibrillation will also be permitted.
9. Patients with another primary malignancy within 3 years prior to starting study treatment with the exception of adequately treated basal cell carcinoma, squamous cell carcinoma or other non-melanomatous skin cancer, or in-situ carcinoma of the uterine cervix.
10. Clinically significant uncontrolled condition(s) including but not limited to: Active uncontrolled infection, Symptomatic congestive heart failure, Unstable angina pectoris or cardiac arrhythmia (subjects with stable atrial fibrillation are not excluded), History of adrenal insufficiency.
11. Psychiatric illness/social situation that would limit compliance with study requirements.
12. Subject has a known infection with HIV, Hepatitis B or Hepatitis C.
13. Subject is known to have poorly controlled diabetes mellitus defined as HbA1c > 7%; subjects with a history of transient glucose intolerance due to corticosteroid administration are allowed in this study if all other inclusion/exclusion criteria are met.
14. Any medical condition which in the opinion of the study investigator places the subject at an unacceptably high risk for toxicities.
15. Subject is unable to swallow or absorb oral tablets normally
16. Female subject who is lactating or pregnant.
17. Subject takes CYP3A Inhibitors/Inducers within 7 days prior to the study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-08-05 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S. Hong, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at the Phase I unit at MD Anderson Cancer Center beginning 08/05/16. Enrollment was closed to new patients on 06/09/21 because of sponsor's decision to stop manufacturing the drug. The trial was terminated on 05/12/22.
Pre-assignment Details: Some patients who consented to join the study were ultimately not treated either because of screen failure or imminent loss of drug supply
Groups:
- Part 1: For evaluation of response rate in patients with cancers harboring CDKN2A deletion or mutation
- Part 2 Tumor-specific Expansion: For evaluation of response rate in a specific tumor type harboring CDKN2A deletion or mutation
Period: Overall Study
Arm/Group | Part 1 | Part 2 Tumor-specific Expansion
Started | 12 | 0
Completed | 0 | 0
Not Completed | 12 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 4 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Screen Failure | 3 | 0

BASELINE CHARACTERISTICS:
Population: Part 2 Tumor-specific expansion (trial was terminated before this part was reached)
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 | Part 2 Tumor-specific Expansion | Total
Number analyzed (Participants) | 12 | 0 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 0 | 7
  >=65 years | 5 | 0 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 5
  Male | 7 | 0 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 0 | 11
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 0 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 0 | 12

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Partial or complete response to ilorasertib
Time Frame: through study completion, maximum 18 months
Population: Patients with tumors harboring CDKN2A deletion or mutation
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 | Part 2 Tumor-specific Expansion
Number analyzed (Participants) | 9 | 0
Participants
  Partial Response | 1 | 0
  Complete Response | 0 | 0

2. Primary Outcome: Efficacy Signal
Description: Selection of specific tumor type where the drug is potentially active for recruitment of additional patients (expansion)
Time Frame: through study completion, maximum 18 months
Population: Patients with tumors harboring CDKN2A deletion or mutation
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 | Part 2 Tumor-specific Expansion
Number analyzed (Participants) | 9 | 0
Participants
  Pancreatic cancer | 1 | 0
  Sarcoma | 3 | 0
  Esophageal | 1 | 0
  GIST | 1 | 0
  Cholangiocarcinoma | 2 | 0
  Oral cancer | 1 | 0

3. Secondary Outcome: Safety and Tolerability
Description: Safety and tolerability of ilorasertib.
Time Frame: through study completion, maximum 18 months'
Population: Patients with tumors harboring CDKN2A deletion or mutation
Measure: Number; unit: events
Arm/Group | Part 1 | Part 2 Tumor-specific Expansion
Number analyzed (Participants) | 9 | 0
events
  Serious adverse events | 5 |
  Other adverse events | 20 |

4. Secondary Outcome: Pharmacodynamic Activity
Description: Assessment of the pharmacodynamic effects of ilorasertib by immunohistochemistry for phospho-histone H3
Time Frame: Cycle 1 Day 1 at up to 72 hours prior to the first dose and 2-4 hours after the second dose
Population: No data was collected
Arm/Group | Part 1 | Part 2 Tumor-specific Expansion
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected after the first dose until end of treatment, death, or loss to follow up, maximum 18 months
Description: Part 2 Tumor-specific expansion (trial was terminated before this part was reached)
Arm/Group | Part 1 | Part 2 Tumor-specific Expansion
All-Cause Mortality (participants affected / at risk) | 1/9 | 0/0
Serious Adverse Events (participants affected / at risk) | 5/9 | 0/0
Other Adverse Events (participants affected / at risk) | 7/9 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 (N=9) | Part 2 Tumor-specific Expansion (N=0)
Sepsis (Infections and infestations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Uncontrolled pain (General disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Cervical stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 (N=9) | Part 2 Tumor-specific Expansion (N=0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Oral mucositis (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Dehydration (General disorders) | 3 | 0
Confusion (Nervous system disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Decreased white count (Blood and lymphatic system disorders) | 1 | 0
AST (Gastrointestinal disorders) | 1 | 0
Bilirubin (Gastrointestinal disorders) | 1 | 0
Knee pain (General disorders) | 1 | 0
Change of skin sensitivity (Skin and subcutaneous tissue disorders) | 1 | 0
Low ANC (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Non-cardiac chest pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-03): https://cdn.clinicaltrials.gov/large-docs/20/NCT02478320/Prot_SAP_000.pdf